CLINICAL TRIAL: NCT00068406
Title: A Phase II Trial of Radiation Therapy and Weekly Cisplatin Chemotherapy for the Treatment of Locally-Advanced Squamous Cell Carcinoma of the Vulva
Brief Title: Chemotherapy, Radiation Therapy, and Surgery in Treating Patients With Locally Advanced Cancer of the Vulva
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0205; NCI-2009-00582 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000322259; GOG-0205 (Other: Gynecologic Oncology Group); GOG-0205 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2011-10

CONDITIONS: Stage III Vulvar Cancer; Stage IVB Vulvar Cancer; Vulvar Squamous Cell Carcinoma
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Radiotherapy, Conformal; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum

ARMS (1):
- Treatment (conventional surgery, radiation therapy, cisplatin) (Experimental): Patients undergo radiotherapy daily on days 1-5 and receive concurrent cisplatin IV over 30 minutes on day 1. Treatment repeats weekly for approximately 6.5 weeks (a total of 32 fractions of radiotherapy) in the absence of unacceptable toxicity.
  Six to eight weeks after the completion of chemoradiotherapy, patients with a complete clinical response may undergo incisional biopsy of the primary tumor and bilateral inguinal/femoral nodes (if the groin nodes were initially unresectable). Patients with microscopic or gross resectable residual disease may then undergo radical resection of the residual tumor. Patients with unresectable disease after the completion of chemoradiotherapy receive additional radiotherapy with 1-2 courses of concurrent cisplatin.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Cisplatin; Procedure: Conventional Surgery

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy
  Other Names: 3-dimensional radiation therapy; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Conventional Surgery

SUMMARY:
This phase II trial is studying how well giving radiation therapy together with cisplatin followed by surgery works in treating patients with locally advanced cancer of the vulva. Drugs used in chemotherapy such as cisplatin use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving chemotherapy with radiation therapy before surgery may shrink the tumor so it can be removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the efficacy of radiotherapy and cisplatin, in terms of achieving a complete clinical and pathological response, in patients with locally advanced squamous cell carcinoma of the vulva that is not amenable to standard radical vulvectomy.

II. Determine the toxicity of this regimen followed by surgery in these patients.

OUTLINE: This is a multicenter study.

Patients undergo radiotherapy daily on days 1-5 and receive concurrent cisplatin IV over 30 minutes on day 1. Treatment repeats weekly for approximately 6.5 weeks (a total of 32 fractions of radiotherapy) in the absence of unacceptable toxicity.

Six to eight weeks after the completion of chemoradiotherapy, patients with a complete clinical response may undergo incisional biopsy of the primary tumor and bilateral inguinal/femoral nodes (if the groin nodes were initially unresectable). Patients with microscopic or gross resectable residual disease may then undergo radical resection of the residual tumor. Patients with unresectable disease after the completion of chemoradiotherapy receive additional radiotherapy with 1-2 courses of concurrent cisplatin.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced squamous cell carcinoma of the vulva

  * T3 or T4 (N0-3, M0)
* Not amenable to surgical resection by standard radical vulvectomy
* Previously untreated disease
* No recurrent disease
* No vulvar melanoma or sarcoma
* Performance status - GOG 0-3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times normal
* Alkaline phosphatase no greater than 3 times normal
* SGOT no greater than 3 times normal
* Creatinine no greater than 2.0 mg/dL
* No gastrointestinal bleeding
* No severe gastrointestinal symptoms
* Capable of tolerating a radical course of chemoradiotherapy
* No septicemia
* No severe infection
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No circumstance that would preclude study completion or follow-up
* No prior cytotoxic chemotherapy
* No prior pelvic radiotherapy
* No concurrent boost brachytherapy
* No prior anticancer therapy that would contraindicate study therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-01; Primary Completion 2010-12 (Actual); Study Completion 2012-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Moore, Principal Investigator — Gynecologic Oncology Group
Locations (103):
- United States (103):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Western Regional CCOP, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Colorado Gynecologic Oncology Group, Aurora, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Rush - Copley Medical Center, Aurora, Illinois
  - University of Illinois, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Gynecologic Oncology of Indiana, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Providence Medical Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Spectrum Health-Blodgett Campus, Grand Rapids, Michigan
  - Gynecologic Oncology of West Michigan PLLC, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Stony Brook University Medical Center, Stony Brook, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates-Midtown, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Knoxville Gynecologic Cancer Specialists PC, Knoxville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Cisplatin + Radiation, Then Surgery: Radiation therapy to the vulva, inguinal-femoral, and lower pelvic lymph nodes by AP-PA fields (180 cGy/daily fraction X 5 days, repeated weekly to a total of 32 fractions- total dose 5760 Gy). Concurrent cisplatin (40 mg/m2) chemotherapy administered weekly throughout radiation therapy. Six to eight weeks following the completion of chemoradiation - surgical excision of gross residual disease in the vulva and/or inguinal-femoral lymph nodes (if the inguinal-femoral nodes were considered unresectable prior to chemoradiation).
Period: Overall Study
Arm/Group | Cisplatin + Radiation, Then Surgery
Started | 61
Completed | 58
Not Completed | 3
Not completed — Ineligible-improper pre-protocol treatm | 1
Not completed — Ineligible-Inadequate Pathology | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Cisplatin + Radiation, Then Surgery
Number analyzed (Participants) | 58
Age, Customized [Count of Participants; unit: Participants]
  Age of participants: <40 years | 5
  Age of participants: 40-49 years | 9
  Age of participants: 50-59 years | 17
  Age of participants: 60-69 years | 13
  Age of participants: >=70 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 54
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Complete Clinical and Pathologic Response
Description: Complete clinical and pathologic response is defined as the disappearance of all gross tumor during chemoradiation with no residual tumor present in the surgical specimen.
Time Frame: Seven weeks after initiating treatment for clinical response and up to fifteen weeks for assessment of pathologic response.
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cisplatin + Radiation, Then Surgery
Number analyzed (Participants) | 58
Percentage of Participants | 50 [39 to 61]

2. Primary Outcome: Treatment-Related Adverse Effects (Grade 3 or Higher) During Study Treatment Period
Description: Number of participants with a maximum grade of 3 or higher during the treatment period. Adverse events are graded and categorized using Common Terminology Criteria for Adverse Events Version 2.0
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment. Up to eleven weeks from the start of study treatment
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin + Radiation, Then Surgery
Number analyzed (Participants) | 58
Participants
  Leukopenia | 18
  Anemia | 4
  Thrombocytopenia | 3
  Neutropenia | 11
  Other Hematologic | 13
  Constitutional | 5
  Cardiovascular | 4
  Dermatologic | 17
  Gastrointestinal | 13
  Genitourinary/Renal | 3
  hemorrhage | 1
  Infection | 8
  Metabolic | 10
  Other Neurologic | 2
  Pulmonary | 1
  Pain | 10
  Sexual/reproductive | 1

ADVERSE EVENTS:
Time Frame: SAE (Serious Adverse Events): All adverse events occurring during study chemo radiation treatment period and up to 30 days after stopping the study treatment are reported without regard to attribution. Up to eleven weeks from the start of study treatment. OAE(Other Adverse Events): All treatment-related adverse events occurring during study chemo radiation treatment period and up to 30 days after stopping the study treatment are reported. Up to eleven weeks from the start of study treatment.
Arm/Group | Cisplatin + Radiation, Then Surgery
Serious Adverse Events (participants affected / at risk) | 17/58
Other Adverse Events (participants affected / at risk) | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin + Radiation, Then Surgery (N=58)
Anemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombosis Embolism (Cardiac disorders) | 2
Ischemia/Cardiac Infarction (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Diarrhea Without Colostomy (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Febrile With Neutropenia (Infections and infestations) | 1
Infection Without Neutropenia (Infections and infestations) | 1
Infection Other (Infections and infestations) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Syncope (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Wound Infectious (Skin and subcutaneous tissue disorders) | 2
Skin Other (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin + Radiation, Then Surgery (N=58)
Leukopenia (Blood and lymphatic system disorders) | 42
Anemia (Blood and lymphatic system disorders) | 51
Thrombocytopenia (Blood and lymphatic system disorders) | 30
Neutropenia (Blood and lymphatic system disorders) | 28
Otherhematologic (Blood and lymphatic system disorders) | 13
Lymphatics (Blood and lymphatic system disorders) | 2
Cardiovascular (Cardiac disorders) | 10
Hearing (Ear and labyrinth disorders) | 3
Endocrine (Endocrine disorders) | 8
Ocular (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 43
Vomiting (Gastrointestinal disorders) | 28
Diarrhea Without Colostomy (Gastrointestinal disorders) | 38
Other Gastrointestinal (Gastrointestinal disorders) | 34
Fatigue (General disorders) | 45
Other Constitutional (General disorders) | 13
Pain Rt (General disorders) | 15
Other Pain (General disorders) | 26
Hepatic (Hepatobiliary disorders) | 6
Allergy (Immune system disorders) | 4
Febrile With Neutropenia (Infections and infestations) | 2
Other Infection (Infections and infestations) | 14
Metabolic (Metabolism and nutrition disorders) | 25
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 4
Neuropathy Motor (Nervous system disorders) | 2
Neuropathy Sensor (Nervous system disorders) | 10
Otherneurologic (Nervous system disorders) | 13
Creatinine (Renal and urinary disorders) | 11
Other Genitourinary/Renal (Renal and urinary disorders) | 21
Vaginal Dryness (Reproductive system and breast disorders) | 3
Other Sexual/Reproductive (Reproductive system and breast disorders) | 3
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 13
Radiation Dermatitis (Skin and subcutaneous tissue disorders) | 11
Rash Desquamation (Skin and subcutaneous tissue disorders) | 29
Wound Not-Infectious (Skin and subcutaneous tissue disorders) | 3
Other Dermatologic (Skin and subcutaneous tissue disorders) | 9
Hemorrhage (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less